CLINICAL TRIAL: NCT06380764
Title: Greater Occipital Nerve Block at Two-levels Spares the Need for Epidural Blood Patch for Management of Postdural Puncture Headache
Brief Title: Greater Occipital Nerve Block Value in Management of Postdural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Yehia Shahin Dabour, Lecturer at Department of Anesthesia, Pain, ICU, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC.11.3.2024
Record Dates: First submitted 2024-04-13; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Blood Patch, Epidural; Saline Solution; Injections; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First line Group (Active Comparator)
  Interventions: Procedure: Greater Occipital Nerve Block; Drug: Lidocaine 2% Injectable Solution
- Second line Group (Active Comparator)
  Interventions: Procedure: Bilateral suboccipital intramuscular injection; Drug: Lidocaine 2% Injectable Solution
- Third line Group (Active Comparator)
  Interventions: Procedure: Epidural Blood Patch
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Normal Saline 10 mL Injection

INTERVENTIONS:
Procedure: Greater Occipital Nerve Block — The occipital artery was localized, while the patient was setting with flexed neck, at the point of meeting of the medial third and the lateral two-thirds of a line drawn extending from the ipsilateral mastoid process to the external occipital protuberance and the GON was located on the medial side of the artery where it exits out of the trapezius fascia into the nuchal line about 5-cm lateral to midline.
  For assurance of GON localization, pressure was applied and the resultant tenderness indicated the site of the nerve. Injection procedure was performed as distal injection at the site of nerve localization and proximal injection was performed at 1.5 cm lateral to the sagittal plane and 3 cm below to the level of the external occipital protuberance.
  Arms: First line Group
Procedure: Bilateral suboccipital intramuscular injection — Sub-occipital intramuscular injection of the prepared solution was carried out on both sides while the patient was setting with maximally flexing the neck to expose these muscles.
  Arms: Second line Group
Procedure: Epidural Blood Patch — Patients showed manifestations of block failure within 24-h after block, received lumbar Epidural blood patch under non-invasive monitoring in the theater. Patient was positioned in the lateral decubitus position, lumbar area was sterilized and the epidural space previously used for receiving the previous neuraxial anesthesia was identified. Fifteen ml of venous blood was obtained aseptically and slowly injected while patient was monitored for the extent of pain severity until complete pain relief.
  Arms: Third line Group
Drug: Normal Saline 10 mL Injection — Placebo drug
  Arms: Placebo Group
Drug: Lidocaine 2% Injectable Solution — Lidocaine is the main drug used in the interventions as it was injected to achieve bilateral block or intramuscular infiltration
  Arms: First line Group; Second line Group

SUMMARY:
Neuraxial techniques are well tolerated and effective options for labor analgesia and anesthesia for caesarean section, and may protect high risk women against severe maternal morbidity. However, neuraxial techniques still have drawbacks especially postdural puncture headache (PDPH) and may be associated with chronic headache, back pain and postnatal depression. PDPH is a relatively common acute complication of neuraxial techniques that was traditionally considered benign and self-limiting, but it significantly impacts patients' general health and quality of life.

Greater Occipital Nerve (GON) originates from C2-3 segments and through its muscular relations it is divided as proximal and distal parts; the most proximal part lies between obliquus capitis inferior and semispinalis and then passes through the semispinalis to pierce the trapezius muscle. In distal region of trapezius fascia, the GON is crossed by the occipital artery and exits the trapezius fascia into the nuchal line about 5-cm lateral to midline. Functionally, GON provides motor supplies to the muscles while passing through it and its main sensory supply is in the occipital region.

ELIGIBILITY:
Inclusion Criteria:

* Patients with postdural puncture headache;
* Patients partially improved on conservative treatment and required a definitive pain relieving management;
* Patients who were intolerant to conventional analgesics;
* Patients who did not receive or did not improve on conservative therapies.

Exclusion Criteria:

* Patients had postdural puncture headache who were improving on conservative treatment and refused further interventions;
* Patients who had headache secondary to local or systemic disease, cervical radiculopathy, manifest diabetes mellitus;
* Patients dependent on routine analgesia for other causes were excluded from the study;
* Patients refused to participate in the study or to sign the written consent;
* Patients missed during follow-up were not included in the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The extent of reduction of consumed analgesia | 7 months
  Necessity of greater occipital nerve block as a management procedure to the postural puncture headache

CONTACTS AND LOCATIONS:
Locations (1):
- Benha university, Banhā, El Qalyoubia, Egypt